CLINICAL TRIAL: NCT03699163
Title: Non-invasive Testing for the Diagnosis and Assessment of Colorectal Disease
Brief Title: The Colorectal Breath Analysis (COBRA) Study
Acronym: COBRA
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial Health Charity (Other); Rosetrees Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17SM3783
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Colorectal Polyps; Colorectal Adenocarcinoma
Keywords: Volatile organic compounds; Mass spectrometry; Early detection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non cancer control patients: Patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure. Those without a finding of colorectal adenocarcinoma will go into this group.
  Interventions: Diagnostic Test: Breath sample
- Colorectal cancer patients: Patients who have known pre-diagnosed colorectal cancer (adenocarcinoma) attending hospital as part of their clinical care will be asked to give a breath sample prior to their cancer operation. Patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure. Those with a finding of colorectal adenocarcinoma will go into this group.
  Interventions: Diagnostic Test: Breath sample

INTERVENTIONS:
Diagnostic Test: Breath sample — Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.

SUMMARY:
This study aims to determine whether a breath test could be used for early detection of colorectal cancer and colorectal polyps.

Patients who are attending for a planned colonoscopy or who are scheduled to undergo elective resection of histologically confirmed colorectal cancer (adenocarcinoma) will be approached to provide a breath sample.

Multi platform mass spectrometry analysis will be performed to establish volatile biomarkers that can discriminate between colorectal cancer, benign colorectal disease (e.g. polyps) and healthy controls.

DETAILED DESCRIPTION:
Colorectal cancer is the 2nd most common cause of cancer death in the UK where survival rates are among the lowest in Europe. If diagnosed early survival may exceed 90%.

The proposed breath test is a non-invasive investigation that can detect the presence of volatile organic compounds (VOCs) in breath and their relative abundance in disease states including colorectal cancer. This test has potential to be used in a primary care setting to identify patients at high risk of colorectal cancer, supporting earlier referral for definitive investigation. A negative test may provide reassurance to patients and prevent unnecessary tests in this group. The test could also have an application for colorectal cancer screening.

In this study the investigators will determine the diagnostic accuracy of an exhaled breath test for the detection of colorectal adenocarcinoma and colonic polyps. To determine the accuracy of the breath test a multicentre cross-sectional study will be conducted to analyse single breath samples from patients attending hospital for planned colonoscopy or elective resection of histologically confirmed colorectal cancer. The target for the study is 1463 patients.

Breath collection will be conducted using a previously validated method. Samples of breath (500ml) collected using a CE-marked handheld ReCIVA sampling device (Owlstone Medical Ltd., Cambridge, UK) during a period of tidal breathing (approximately 5minutes) will be absorbed onto thermal desorption tubes (Markes International, Llantrisant, UK). All patients will have received bowel preparation and will be fasted for a minimum of 6 hours prior to the breath sample. Breath samples collected within thermal desorption tubes will be transferred to a central laboratory for analysis by gas chromatography mass spectrometry (GC-MS) and proton transfer reaction time of flight mass spectrometry (PTR-ToF-MS). Raw data files will be extracted and analysed in accordance with established protocols. Quality assurance measures will be formally assessed at each stage of sample handling.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and ≤90 years of age
* Undergoing planned colonoscopy or elective resection of histologically confirmed colorectal adenocarcinoma
* Fasted >6 hours
* Able to provide informed written consent

Exclusion Criteria:

* Any patient <18 years or >90 years of age.
* Lacks capacity or is unable to provide informed written consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are attending for a planned colonoscopy or who are scheduled to undergo elective resection of histologically confirmed colorectal adenocarcinoma will be eligible for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 1855 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George B Hanna, FRCS PhD, Principal Investigator — Imperial College London
Locations (8):
- United Kingdom (8):
  - Homerton Hospital, London
  - St Mark's Hospital, London
  - St George's Hospital, London
  - Chelsea and Westminster Hospital, London
  - Royal Marsden Hospital, London
  - West Middlesex Hospital, London
  - St Mary's Hospital, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Woodfield G, Belluomo I, Laponogov I, Veselkov K; COBRA1 WORKING GROUP; Cross AJ, Hanna GB. Diagnostic Performance of a Noninvasive Breath Test for Colorectal Cancer: COBRA1 Study. Gastroenterology. 2022 Nov;163(5):1447-1449.e8. doi: 10.1053/j.gastro.2022.06.084. Epub 2022 Jul 5. No abstract available. PMID 35803311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1855 total patients were enrolled in the study between 5/6/2017 and 21/2/2020.
Pre-assignment Details: The cancer/non cancer diagnosis was not known for the majority of excluded participants, because the exclusion was based upon data corruption/failure of quality control of breath sample, hence no further clinical details were recorded. Exclusions have been arbitrarily divided between both study groups for the purposes of this table.
Groups:
- Non-cancer Control Patients: Patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure. Those without a finding of colorectal adenocarcinoma will enter this group.
  Breath sample: Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.
- Colorectal Cancer Patients: Patients who have known pre-diagnosed colorectal cancer (adenocarcinoma) attending hospital as part of their clinical care will be asked to give a breath sample prior to their cancer operation. Patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure. Those with a finding of colorectal adenocarcinoma will enter this group.
  Breath sample: Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.
Period: Overall Study
Arm/Group | Non-cancer Control Patients | Colorectal Cancer Patients
Started | 1487 | 368
Completed | 1270 | 162
Not Completed | 217 | 206
Not completed — Physician Decision | 12 | 0
Not completed — failed QC measures | 205 | 206

BASELINE CHARACTERISTICS:
Groups:
- Colorectal Cancer: 162 patients of the included total had a diagnosis of colorectal cancer
- Non-cancer Controls: 1270 patients had a non-cancer diagnosis
- Total: Total of all reporting groups
Arm/Group | Colorectal Cancer | Non-cancer Controls | Total
Number analyzed (Participants) | 162 | 1270 | 1432
Age, Continuous [Median (Full Range); unit: years] | 66.5 [30 to 90] | 63 [18 to 87] | 64 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 540 | 601
  Male | 101 | 730 | 831
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arab | 5 | 40 | 45
  Asian/Asian British | 22 | 198 | 220
  Black / African / Caribbean / Black British | 19 | 106 | 125
  Other ethnicity | 8 | 38 | 46
  Unrecorded | 4 | 30 | 34
  White British/ European | 104 | 858 | 962
Time fasted [Median (Full Range); unit: Hours] | 22 [4 to 36] | 24 [7 to 72] | 24 [4 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Determine the Diagnostic Accuracy of the Proposed Breath Test for Detection of Colorectal Cancer in All Patients
Description: Diagnostic accuracy will be measured by calculating the sensitivity and specificity of the test for detection of colorectal cancer, as diagnosed on colonoscopy, using 14 specific VOCs plus BMI as prediction variables.
Time Frame: 30 minutes
Measure: Number; unit: percentage of true cases
Groups:
- Detection of Colorectal Cancer in Breath in All Patients: Colorectal cancer patients attending for surgery and non-cancer controls attending for colonoscopy
Arm/Group | Detection of Colorectal Cancer in Breath in All Patients
Number analyzed (Participants) | 1432
percentage of true cases
  Sensitivity | 79
  Specificity | 86

2. Primary Outcome: Determine the Diagnostic Accuracy of Using VOCs Present in Breath for the Detection of Colorectal Cancer in Symptomatic Patients
Description: as for outcome 1
Time Frame: 30 minutes
Population: This a subgroup or 855 symptomatic patients taken from within the total cohort
Measure: Number; unit: Percentage of true cases
Groups:
- Detection of Colorectal Cancer in Breath in Symptomatic Patients: Symptomatic patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure. Those with no finding of colorectal adenocarcinoma entered this group.
  Breath sample: Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.
Arm/Group | Detection of Colorectal Cancer in Breath in Symptomatic Patients
Number analyzed (Participants) | 855
Percentage of true cases
  Sensitivity | 83
  Specificity | 88

ADVERSE EVENTS:
Time Frame: 30 minutes
Description: Any report of any adverse event/symptom/experience relating to the breath testing process, from any patient
Groups:
- Endoscopy Patients: Patients who are attending hospital for a colonoscopy as part of their routine clinical care, or as part of the Bowel Cancer Screening Programme, will be asked to give a sample of their breath prior to the procedure.
  Breath sample: Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.
- Colorectal Cancer Patients: Patients who have known pre-diagnosed colorectal cancer (adenocarcinoma) attending hospital as part of their clinical care will be asked to give a breath sample prior to their cancer operation.
  Breath sample: Patients will be asked to give a sample of their breath, using the ReCIVA breath testing device. This involves performing tidal breathing whilst wearing a face mask for approximately 5 minutes. Breath (500mls at a flow rate of 200mls/min) is passed over thermal desorption tubes which absorb compounds of interest.
Arm/Group | Endoscopy Patients | Colorectal Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/1270 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/1270 | 0/162
Other Adverse Events (participants affected / at risk) | 0/1270 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03699163/Prot_SAP_000.pdf